CLINICAL TRIAL: NCT06383572
Title: Phase I/II Study of Engineered T Cell Receptor-Modified NK Cells Targeting PRAME in Conjunction With Lymphodepleting Chemotherapy for the Management of Relapse/Refractory Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0196; NCI-2024-03505 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lymphodepleting Chemotherapy; Myeloid Malignancies
MeSH Terms: interventions — Cyclophosphamide; fludarabine phosphate; fludarabine; Decitabine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 (Dose Escalation and Dose Expansion) (Experimental): Participants will be assigned to a dose level of the NK cell treatment based on when you join this study. Up to 4 dose levels of the treatment will be tested.
  The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the NK cell treatment is found.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine phosphate; Drug: Decitabine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclophosphamide — Given by IV
  Other Names: Cytoxan®; Neosar®
Drug: Fludarabine phosphate — Given by IV
  Other Names: Fludarabine; Fludara®
Drug: Decitabine — Given by IV
  Other Names: Dacogen
Drug: Dexamethasone — Given by mouth
  Other Names: Decadron

SUMMARY:
To find a recommended dose of PRAME-TCR-NK cells that can be given to patients with AML or MDS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess dose-limiting toxicity (DLT) and determine the safety, day 30 response rate, day 180 treatment failure rate (defined as disease progression or death) and optimal cell dose of T cell receptor (TCR) modified cord blood-natural killer (CB-NK) cells (TCR-NK) targeting PRAME in patients with relapsed/refractory myeloid malignances, for each of the following diseases; AML, and MDS/CMML. The day 30 response rate and day 180 treatment failure rate will be estimated, and the estimates will be used to identify an optimal dose of PRAME-TCR-NK cells.

SECONDARY OBJECTIVES:

I. To assess the preliminary efficacy of PRAME-TCR-NK cells (day+ 30 complete and partial response rates; day 180 progression-free survival rate) in patients with relapsed/refractory AML and MDS.

II. To quantify persistence of infused allogeneic donor PRAME-TCR CB-derived NK cells in the recipient as an integrated evaluation.

III. To conduct comprehensive immune reconstitution studies.

IV. To obtain preliminary data on quality of life and patient experience (Patient Reported Outcomes Measurement Information Systems [PROMIS]-29 quality of life questionnaire score).

OUTLINE:

This is a phase I dose-escalation study of PRAME-TCR-NK followed by a phase II study.

Patients receive dexamethasone orally (PO) on days -10, -9, -8, -7, and -6, decitabine intravenously (IV) over 1 hour on days -6, -5, and -4, fludarabine IV over 30 minutes and cyclophosphamide IV over 60 minutes on days -5, -4, and -3 and PRAME-TCR-NK cells IV over 2-20 minutes on day 0. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) and computed tomography (CT) or chest x-ray pre-treatment and bone marrow aspiration and biopsy, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up for 24 months then for at least 15 years per protocol PA17-0483.

Sponsor: M D Anderson Cancer Center

Lead Organization: M D Anderson Cancer Center

Principal Investigator: Ramdial, Jeremy

Responsible Party: Sponsor

Overall Official: Ramdial, Jeremy (Principal Investigator), M D Anderson Cancer Center

ELIGIBILITY:
Inclusion Criteria:

1. 18- 80 years of age. English and non-English speaking patients are eligible.
2. Patients with one of the following hematological malignances: AML, MDS/CMML. Patients must meet disease specific eligibility criteria (see below)
3. Patients at least 7 days from last cytotoxic chemotherapy at the time of starting lymphodepleting chemotherapy, except for Hydroxyurea which is allowed for peripheral blood count control in AML patients until the day prior to administration of lymphodepleting chemotherapy. Patients may continue tyrosine kinase inhibitors or other targeted therapies until up to three days prior to administration of lymphodepleting chemotherapy.
4. Localized radiotherapy to one or more disease sites is allowed prior the infusion provided that there are additional disease sites that are not irradiated to assess response.
5. Karnofsky Performance Scale > 50%.
6. Adequate organ function: as described in 7-10
7. Renal: Serum creatinine </= 2.0 mg/dL and estimated Glomerular Filtration Rate (eGFR using the CKD-EPI equation).GFR = 141 x [min(Scr/k), 1)a x max (Scr/k), 1) -1.209] x Age-0.993 x 1.018 [if female] x [ 1.157 if Black] (a is 0.329 for females and 0.411 for males; min indicates minimum of Scr/k or 1, and max indicates maximum of Scr/k or 1)
8. Hepatic: ALT/AST </= 2.5 x ULN or </= 5 x ULN if documented liver metastases, Total bilirubin </= 1.5 mg/dL, except in subjects with Gilbert's Syndrome in whom total bilirubin must be </= 3.0 mg/dL. No history of liver cirrhosis. No ascites.
9. Cardiac: Cardiac ejection fraction >/= 40%, no clinically significant pericardial effusion as determined by an ECHO/MUGA, and no uncontrolled arrhythmias or symptomatic cardiac disease.
10. Pulmonary: No clinically significant pleural effusion (per PI discretion), baseline oxygen saturation > 92% on room air and adequate pulmonary function with FEV1, FVC and DLCO (corrected for Hgb) >50%.
11. Able to provide written informed consent.
12. All participants who are able to have children must practice effective birth control while on study and up to 3 months post completion of study therapy. Acceptable forms of birth control for female patients include: hormonal birth control, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence, for the length of the study. If the participant is a female and becomes pregnant or suspects pregnancy, she must immediately notify her doctor. If the participant becomes pregnant during this study, she will be taken off this study.

    a. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physicaian immediately.
13. Men treated or enrolled on this protocol must also agree to use adequate contraception, such as subject post vasectomy, partner with implantable or oninjectable contraceptives, and condoms plus spermicide, prior to the study, for the duration of study participation, and 4 months after completion of study agent administration. Men who are able to have children must use effective birth control while on the study. If the male participant fathers a child or suspects that he has fathered a child while on the study, he must immediately notify his doctor.
14. Signed consent to long-term follow-up protocol PA17-0483 to fulfill the institutional responsibilities to various regulatory agencies.
15. Life Expectancy >=3 mo, by PI assessment
16. Patients are HLA-A*02:01 positive on HLA typing.
17. Patients must have one of the following diseases:

Acute myeloid leukemia (AML): one of the following:

1. Patients with active (>5% of blasts or positive MRD at a level of >0.1% measured by multiparameter flow cytometry) relapsed or refractory AML. Who have received at least two lines of therapy. One or more of the lines of therapy must include hypomethylating agents and venetoclax. Patients who have mutations for which there are FDA approved targeted therapies (i.e. FLT3) must also have received at least one of such agent. Patients with diagnosis of acute promyelocytic leukemia are not eligible. Patients who relapse after allogeneic stem cell transplantation are eligible irrespective of the number and type of therapy received prior transplant.

1. Relapsed AML is defined as patients who had a first complete remission (CR) before developing recurrent disease.
2. Refractory AML is defined as patients that have not achieved a CR after 2 cycles of standard induction chemotherapy.

OR determining the eligibility of the patient. For example, patients who received hypomethylating agents and venetoclax for the treatment of the MDS are not required to receive again hypomethylating agents and venetoclax to treat the secondary AML to be eligible. Similarly, patients who received two lines of therapy for the management of the MDS or MPD are not required to receive an additional two lines of therapy for the management of the AML to be eligible. Patients who relapse after allogeneic stem cell transplantation are eligible irrespective of the number and type of therapy received prior transplant.

Myelodysplastic syndromes (MDS)/Chronic myelomonocytic leukemia (CMML):one of the following:

1. Patients with high risk or intermediate risk MDS/CMML who have received at least two lines of therapy and have positive MRD at a level of >0.1% measured by multiparameter flow cytometry or are not in morphological remission.

   OR
2. Patients with relapse high risk or intermediate risk MDS/CMML after at least 2 lines of therapy. Relapse is defined as positive MRD at a level of >0.1% measured by multiparameter flow cytometry or loss of morphological remission.

   OR
3. CMML patients with refractory disease defined as failure to achieve complete remission after 4 therapy cycles of hypomethylating agent therapy or relapse or progression after any number of cycles of therapy.
4. Patients with MDS/CMML who relapse after allogeneic stem cell transplantation are eligible irrespective of the number and type of therapy received prior to transplant.

Exclusion Criteria:

1. Positive beta HCG in female of child-bearing potential defined as not postmenopausal for 24 months or no previous surgical sterilization or lactating females.
2. Presence of clinically significant Grade 3 or greater toxicity from the previous treatment, as determined by PI.
3. Presence of uncontrolled fungal, bacterial, viral, or other infection not responding to appropriate therapy.
4. Known active hepatitis B or C.
5. Known HIV with detectable viral load
6. Presence of active neurological disorder(s).
7. Active autoimmune disease within 12 months of enrollment
8. Active cerebral or meningeal involvement by the malignancy
9. Active (defined as requiring therapy) acute or chronic GVHD
10. Any other malignancy known to be active, except for treated cervical intra-epithelial neoplasia and non-melanoma skin cancer.
11. Presence of any other serious medical condition that may endanger the patient at investigator discretion.
12. Major surgery <4 weeks prior to first dose of the preparatory chemotherapy
13. Allogeneic SCT or DLI <12 weeks prior to first dose of preparatory chemotherapy
14. Concomitant use of other investigational agents.
15. Concomitant use of other anti-cancer agents.
16. Patients receiving systemic steroid therapy at time of enrollment (physiological substitutive doses deemed per PI assessment are allowed),or have received antithymocyte globulin or lymphocyte immune globulin within 14 days of enrollment or alemtuzumab within 28 days of enrollment.
17. Patients receiving immunosuppressive therapy such as steroids and calcineurin inhibitors.

Criteria to Receive Lymphodepletion Chemotherapy:

Within 72 hours prior to the start of Lymphodepletion chemotherapy, subjects must meet the eligibility criteria outlined below:

1. No uncontrolled active systemic infection. Subjects must be fever free for at least 48 hours without antipyretics unless the patient is felt to have tumor fever.
2. Absence of clinically significant Grade 3 or greater toxicity from the previous treatment, as determined by the Principal Investigator.
3. Patient should not be receiving systemic steroids above physiologic dosing (excluding dexamethasone 25mg/m^2 PO as noted in the treatment plan from Day -10 through Day -6.) or calcineurin inhibitors.
4. Patients should be at least 7 days from last cytotoxic chemotherapy at the time of starting lymphodepleting chemotherapy, except for Hydroxyurea which is allowed for peripheral blood count control in AML patients until the day prior to administration of lymphodepleting chemotherapy.
5. Patients may continue tyrosine kinase inhibitors or other targeted therapies until up to three days prior to administration of lymphodepleting chemotherapy

Criteria Prior to NK Cell Infusion:

On Day 0, prior to the NK Cell infusion, subjects must meet the eligibility criteria for infusion outlined

1. No active and uncontrolled systemic infection. Subjects must be fever free for 48 hours without antipyretic unless patient is felt to have tumor fever.
2. No clinical signs of cardiac failure.
3. Oxygen saturation levels (SPO2) >92%
4. No other ongoing medical condition that in the opinion of the investigator can affect patient's safety.
5. No rapidly progressing AML/MDS.
6. Patient must be able to be off of all steroid treatment within 24hrs of cell infusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Ramdial, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org